CLINICAL TRIAL: NCT04503824
Title: Assessing LncRNA DQ786243 and IL-17 Expression in Oral Lichen Planus: A Case Control Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Mahmoud Abdel Wahed Abdel dayem, assistant lecterur, Cairo University
Other Study IDs: 14422019590827
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Patients With Oral Lichen Planus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group IIa: 13 papular OLP
  Interventions: Diagnostic Test: saliva samples
- Group IIb: 13 atrophic OLP
  Interventions: Diagnostic Test: saliva samples
- Group IIc: 13 erosive OLP
  Interventions: Diagnostic Test: saliva samples
- Group I: 13 healthy individuals
  Interventions: Diagnostic Test: saliva samples

INTERVENTIONS:
Diagnostic Test: saliva samples — Salivary expression of lncRNA DQ786243 and IL-17 will be evaluated using qRT-PCR.

SUMMARY:
Observational case-control study. The current study aims to assess the salivary expression of lncRNA DQ786243 and IL-17 in OLP, to better understand the pathogenesis of OLP and provide effective targets for OLP therapy.

DETAILED DESCRIPTION:
Oral lichen planus (OLP) is a common chronic inflammatory disease associated with cell-mediated immunological dysfunction. OLP can be seen in different clinical presentations. It can be classified as papular (reticular), atrophic (erythematous) and erosive (ulcerative, bullous).1 Numerous predisposing factors have been blamed for causing OLP, including: stress, diabetes, drugs, dental materials, autoimmune diseases, infectious agents and genetic predisposition. 2 Regarding the pathogenesis of OLP, it is a T-cell mediated inflammatory disease where antigen- specific and non-specific mechanisms are hypothesized to be involved3. Antigen-specific mechanisms include antigen presentation by basal keratinocytes and antigen-specific keratinocyte killing by CD8+ cytotoxic T-cells. Non-specific mechanisms include mast cell degranulation, basement membrane disruption, chemokines and matrix metalloproteinase (MMP) activation in OLP lesions.4 Various treatment regimens have been proposed to improve the management of symptomatic OLP, but a permanent cure is not yet available. Treatment regimens are non-specific and directed at eliminating inflammation and immunosuppression.5 Corticosteroids constitute the main stay agent, other available treatment modalities include immunosuppressants, cyclosporin, tacrolimus, and retinoids.6 Long non-coding RNAs (lncRNAs) have been identified as new regulatory molecules. They modulate protein coding gene at the chromatin remodeling level, or the transcriptional and post- transcriptional control level. They play vital roles in cell differentiation, cell growth and apoptosis. lncRNA DQ786243 is drawing attention in the pathogenesis of a variety of inflammatory immune- mediated diseases such as Crohn's disease and OLP.7, 8 A recent study suggested that lncRNA DQ786243 exert its function through interleukins (ILs) including IL-17. T-helper 17 response and its hallmark IL-17 is gaining more evidence for its role and association with many diseases such as

5 Crohn's disease, ulcerative colitis, systemic lupus erythematosus and OLP. IL-17 has been found to participate in the development of autoimmune disease, inflammatory destruction and tumor microenvironments.9, 10

Research question:

What is the salivary expression of lncRNA DQ786243 and IL-17 in Oral Lichen Planus? Population (P): Oral lichen planus Control (C): Healthy individuals Outcome (O): Salivary expression level of lncRNA DQ786243 and IL-17

Objectives:

The current study aims to assess the salivary expression of lncRNA DQ786243 and IL-17 in OLP, to better understand the pathogenesis of OLP and provide effective targets for OLP therapy.

III. Methods:

7. Study design Observational case-control study. 8. Settings Participants will be recruited from the diagnostic centre and Oral Medicine clinic of the Faculty of Dentistry- Cairo University. The recruitment period is expected to extend from January 2020 to January 2021.

A) Participants 9. Eligibility criteria

Inclusion criteria:

* Patients diagnosed with OLP.
* Patient who will agree to participate in the study.
* Patients who will accept to sign the informed consent.

Exclusion criteria:

* Patients suffering from any systemic disease.
* Patients suffering from any local inflammatory disease or infection.
* Pregnant and lactating women. ▪ Smokers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with OLP.

  * Patient who will agree to participate in the study.
  * Patients who will accept to sign the informed consent.

Exclusion Criteria:

* Patients suffering from any systemic disease.

  * Patients suffering from any local inflammatory disease or infection.
  * Pregnant and lactating women. ▪ Smokers.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: thestudy composes of two groups: healthy controls and OLP. The expression of the two markers will be compared between the two studied groups. In OLP group, the expression of the two markers will be correlated with pain and clinical assessment scores. In addition, OLP group will be subgrouped based on the clinical form: papular, atrophic, erosive. Data of all participants will be entered on Excel sheet. Each participant will be provided an ID number that will be used for data management and placed as a label for the samples.
  Group I: 13 healthy individuals Group IIa: 13 papular OLP Group IIb: 13 atrophic OLP Group IIc: 13 erosive OLP
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2021-06-29 (Estimated); Study Completion 2021-07-29 (Estimated)

PRIMARY OUTCOMES:
Salivary expression of lncRNA DQ786243. Salivary expression of lncRNA DQ786243. Salivary expression of lncRNA DQ786243. Salivary expression of lncRNA DQ786243. ▪ Salivary expression of IL-17 and Salivary expression of lncRNA DQ786243. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abdeldayem E, Rashed L, Ali S. Salivary expression of lncRNA DQ786243 and IL-17 in oral lichen planus: case-control study. BMC Oral Health. 2022 Jun 18;22(1):240. doi: 10.1186/s12903-022-02277-0. PMID 35717182